CLINICAL TRIAL: NCT05823025
Title: Withings Study to Analyze the Accuracy of Pulse Wave Velocity Measurement With Bathroom Scales
Brief Title: Withings Study to Analyze the Accuracy of Pulse Wave Velocity Measurement With Bathroom Scales (WIVOP-Scales)
Acronym: WIVOP-Scales
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Withings (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-A00776-37
Record Dates: First submitted 2023-03-24; First posted 2023-04-21 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Vascular Stiffness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypertension: Hypertensive patient
  Interventions: Other: PWV measurement
- Sleep apnea or COPD: Patient having sleep apnea or COPD (Chronic obstructive pulmonary disease)
  Interventions: Other: PWV measurement

INTERVENTIONS:
Other: PWV measurement — Patient will have its PWV measured with the reference (the SphygmoCor) and by stepping on Withings bathroom scales WBS08 and WBS12.

SUMMARY:
The aim of this study is to evaluate the diagnostic performance of Withings bathroom scales WBS08 and WBS12 to measure PWV (Pulse Wave Velocity).

DETAILED DESCRIPTION:
Patients likely to have a high PWV (having hypertension, sleep apnea or chronic obstructive pulmonary disease) are included in hospitals. Each patient will have his PWV measured with Withings WBS08 and WBS12 and its reference the SphygmoCor CvMS.

ELIGIBILITY:
Inclusion Criteria:

* The subject is an adult, man or woman (18 years old or more),
* Subjects affiliated or eligible to a social security system,
* Subjects having expressed their consent to take part in the study.
* Two subsets of patients will be included in the study :

  * Hypertensive patient
  * Patient having sleep apnea or COPD (Chronic obstructive pulmonary disease)

Exclusion Criteria:

* Minors under 18 years old,
* Subject is pregnant,
* Subjects having a pacemaker or an ICD (Implantable cardioverter defibrillator),
* Subjects having refused to give their consent,
* Vulnerable subjects according to the French regulation in force:

  * Individuals deprived of liberty by a court, medical or administrative order,
  * Individuals legally protected or unable to express their consent to take part in the study,
  * Individuals unaffiliated to or not beneficiary of a social security system,
  * Individuals who fit in multiple categories above,
* Individuals linguistically or mentally unable to express their consent,
* Individuals having a lower limb amputation bigger than toes,
* Individuals not able to stand still for a few minutes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient have chronic disease (hypertension, sleep apnea, BPCO) likely to have a high PWV.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Estimated)
Dates: Start 2023-05-02 (Estimated); Primary Completion 2024-05-02 (Estimated); Study Completion 2024-11-02 (Estimated)

PRIMARY OUTCOMES:
PWV measurement bias | 1 year
  Difference between the PWV measured and the PWV reference (m.s-1)
PWV measurement deviation | 1 year
  The standard deviation of the difference between the PWV measured and the PWV reference (m.s-1)

SECONDARY OUTCOMES:
Safety use | 1 year
  The percentage of participant having adverse effects over the total number of participant included.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Boutouyrie, Pr, Principal Investigator — Georges Pompidou european hospital
Locations (2):
- France (2):
  - CHU Grenoble, Grenoble, Auvergne-Rhône-Alpes
  - Georges Pompidou European Hospital, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No